CLINICAL TRIAL: NCT00296504
Title: An Open-Label Phase III Study to Assess the Long Term Safety Profile of GW433908 Containing Regimens in HIV-1 Infected Subjects
Brief Title: A Study To Assess GW433908 (Fosamprenavir) Containing Regimens In HIV-1 Infected Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: APV30005
Record Dates: First submitted 2006-02-24; First posted 2006-02-27 (Estimated); Results first posted 2011-11-08 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2012-06

CONDITIONS: Infection, Human Immunodeficiency Virus
Keywords: antiretroviral therapy naive subjects; fosamprenavir; HIV-1; protease inhibitor; pro-drug; antiretroviral therapy; LEXIVA; AGENERASE; GW433908; amprenavir
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — fosamprenavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: fosamprenavir (GW433908)
Drug: ritonavir
  Other Names: fosamprenavir (GW433908)

SUMMARY:
GW433908 (fosamprenavir; FPV)is a pro-drug of amprenavir (APV) which is more water soluble and can be formulated into a tablet with a reduced pill burden (four 700mg tablets of FPV versus sixteen 150mg capsules daily for APV. This study is designed to provide additional information on long term safety and tolerability of FPV containing regimens for those subjects who received FPV in previous GlaxoSmithKline studies.

DETAILED DESCRIPTION:
ViiV Healthcare is the new sponsor of this study, and GlaxoSmithKline is in the process of updating systems to reflect the change in sponsorship.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant/non-lactating females >/=13 years of age (or >/= 18 years of age according to local requirements).
* Received fosamprenavir through prior participation in APV20001, APV30002, APV30003 or PRO30017 or have participated in APV30001 or other studies as deemed appropriate by the project team.

Exclusion Criteria:

* Permanent discontinuation of GW433908 in a previous study due to intolerance.
* An active CDC Class C Event.
* Any condition which, in the opinion of the investigator, would preclude a subject from participation.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 753 (Actual)
Dates: Start 2001-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (21):
- United States (9):
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Manhasset, New York
  - GSK Investigational Site, Galveston, Texas
- GSK Investigational Site, Campinas, São Paulo, Brazil
- GSK Investigational Site, Santiago, Región Metro de Santiago, Chile
- France (5):
  - GSK Investigational Site, Le Kremlin-Bicêtre
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Vandœuvre-lès-Nancy
  - GSK Investigational Site, Villejuif
- GSK Investigational Site, Genoa, Liguria, Italy
- GSK Investigational Site, Coimbra, Portugal
- Spain (2):
  - GSK Investigational Site, Badajoz
  - GSK Investigational Site, Barcelona
- GSK Investigational Site, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: APV30005 enabled Human Immunodeficiency Virus (HIV)-infected participants who had received a Fosamprenavir (FPV)-containing or other regimen in a number of studies, including APV30001, APV30002, and APV30003, to receive FPV until 31 January 2006 (Interim Analysis) or until commercial supplies of FPV were available locally, whichever was later.
Pre-assignment Details: Participants are divided into arms depending on the regimen they received in Studies APV30001, APV30002, and APV30003 or whether they were PI-naïve or PI-experienced at the time they enrolled into other studies. For the final analysis, 111 participants are included who continued in APV30005 after 31 January 2006 until study completion.
Groups:
- FPV Population (APV30001): Fosamprenavir (FPV) +/- ritonavir (RTV) + background regimen in participants who had received FPV in APV30001 (NCT00008554)
- NFV Population (APV30001): FPV +/- RTV + background regimen in participants who had received nelfinavir (NFV) in APV30001
- FPV Population (APV30002): FPV +/- RTV + background regimen in participants who had received FPV in APV30002 (NCT00009061)
- NFV Population (APV30002): FPV +/- RTV + background regimen in participants who had received NFV in APV30002
- FPV/RTV Once Daily (QD) Population (APV30003): FPV +/- RTV + background regimen in participants who had received FPV/RTV QD in APV30003 (no NCT number)
- FPV/RTV Twice Daily (BID) Population (APV30003): FPV +/- RTV + background regimen in participants who had received FPV/RTV BID in APV30003
- Protease Inhibitor (PI)-Naïve Population (Other Studies): FPV +/- RTV + background regimen in participants who were PI-naïve prior to enrollment in the parent study
- PI-Experienced Population (Other Studies): FPV +/- RTV + background regimen in participants who were PI-experienced prior to enrollment in the parent study
- Final Analysis Population (APV30005): FPV +/- RTV + background regimen in participants who remained in APV30005 after 31 January 2006
Period: Interim Analysis
Arm/Group | FPV Population (APV30001) | NFV Population (APV30001) | FPV Population (APV30002) | NFV Population (APV30002) | FPV/RTV Once Daily (QD) Population (APV30003) | FPV/RTV Twice Daily (BID) Population (APV30003) | Protease Inhibitor (PI)-Naïve Population (Other Studies) | PI-Experienced Population (Other Studies) | Final Analysis Population (APV30005)
Started | 119 | 18 | 221 | 54 | 73 | 78 | 104 | 86 | 0
Ongoing | 32 | 12 | 16 | 22 | 0 | 0 | 30 | 1 | 0
Completed | 43 | 0 | 116 | 11 | 36 | 41 | 30 | 37 | 0
Not Completed | 76 | 18 | 105 | 43 | 37 | 37 | 74 | 49 | 0
Not completed — Withdrawal by Subject | 8 | 0 | 12 | 0 | 5 | 5 | 9 | 3 | 0
Not completed — Lost to Follow-up | 13 | 3 | 26 | 8 | 14 | 4 | 11 | 4 | 0
Not completed — Clinical Progression | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 2 | 0
Not completed — Insufficient Viral Load Response | 5 | 1 | 12 | 2 | 7 | 9 | 2 | 24 | 0
Not completed — Adverse Event | 0 | 0 | 13 | 4 | 6 | 3 | 4 | 5 | 0
Not completed — Protocol Violation | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Insufficient CD4 Response | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Not completed — Switched to Commercially Available Drug | 2 | 0 | 4 | 1 | 0 | 5 | 3 | 4 | 0
Not completed — Pregnancy | 4 | 1 | 4 | 2 | 0 | 1 | 1 | 1 | 0
Not completed — Death | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participant Non-compliant | 0 | 1 | 2 | 1 | 1 | 3 | 6 | 2 | 0
Not completed — Participant Wanted to Become Pregnant | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — To Simplify Treatment | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Participant Had Problems with Alcohol | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Participant Moved | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0
Not completed — Participant Was Incarcerated | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Resistance to FPV | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Principle Investigator Discretion | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Principle Investigator Terminated Study | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-adherence | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Site Closing | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Not completed — Lack of Personnel at Site | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Missed Schedule Date | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Inclusion in Other Protocol | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Participant Stopped | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician and Participant Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Participant Stopped HIV Medications | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Study Ended | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Participant Needed Interferon | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Ongoing | 32 | 12 | 16 | 22 | 0 | 0 | 30 | 1 | 0
Period: Final Analysis
Arm/Group | FPV Population (APV30001) | NFV Population (APV30001) | FPV Population (APV30002) | NFV Population (APV30002) | FPV/RTV Once Daily (QD) Population (APV30003) | FPV/RTV Twice Daily (BID) Population (APV30003) | Protease Inhibitor (PI)-Naïve Population (Other Studies) | PI-Experienced Population (Other Studies) | Final Analysis Population (APV30005)
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 111 (Continued in study; commercial supplies of FPV were unavailable locally at end of Interim Analysis.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 90
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 21
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5
Not completed — Insufficient Viral Load Response | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Not completed — Tuberculosis | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Participant Moved to Another Country | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Poor Adherence | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- FPV Population (APV30001): FPV +/- RTV + background regimen in participants who had received FPV in APV30001 (NCT00008554)
- NFV Population (APV30001): FPV +/- RTV + background regimen in participants who had received NFV in APV30001
- FPV/RTV QD Population (APV30003): FPV +/- RTV + background regimen in participants who had received FPV/RTV QD in APV30003 (no NCT number)
- FPV/RTV BID Population (APV30003): FPV +/- RTV + background regimen in participants who had received FPV/RTV BID in APV30003
- PI-Naïve Population (Other Studies): FPV +/- RTV + background regimen in participants who were PI-naïve prior to enrollment in the parent study
- Total: Total of all reporting groups
Arm/Group | FPV Population (APV30001) | NFV Population (APV30001) | FPV Population (APV30002) | NFV Population (APV30002) | FPV/RTV QD Population (APV30003) | FPV/RTV BID Population (APV30003) | PI-Naïve Population (Other Studies) | PI-Experienced Population (Other Studies) | Total
Number analyzed (Participants) | 119 | 18 | 221 | 54 | 73 | 78 | 104 | 86 | 753
Age, Customized [Mean (Full Range); unit: years] | 36.3 [17 to 70] | 35.8 [22 to 54] | 37.7 [19 to 69] | 36.2 [26 to 63] | 41.9 [27 to 58] | 42.3 [24 to 71] | 39.3 [21 to 75] | 40.2 [19 to 60] | 38.7 [17 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 9 | 63 | 23 | 9 | 12 | 24 | 22 | 198
  Male | 83 | 9 | 158 | 31 | 64 | 66 | 80 | 64 | 555
Race/Ethnicity, Customized [Number; unit: participants]
  White | 34 | 1 | 109 | 14 | 59 | 56 | 44 | 77 | 394
  Black | 35 | 6 | 86 | 34 | 10 | 14 | 34 | 7 | 226
  Asian | 1 | 0 | 4 | 0 | 1 | 1 | 1 | 0 | 8
  American Hispanic | 49 | 11 | 16 | 2 | 3 | 7 | 23 | 2 | 113
  Other: Race Not Specified | 0 | 0 | 6 | 4 | 0 | 0 | 2 | 0 | 12
Number of Participants with the Indicated CDC Classification of HIV Infection [Number; unit: participants] — The Centers for Disease Control and Prevention (CDC) 1993 classification system for HIV infection was based on three clinical categories (A, B, and C). Category A comprised asymptomatic acute or primary HIV infection or persistent generalized lymphadenopathy (lymphnode disease). Category B comprised symptomatic conditions not included in clinical categories A or C but attributed to a cell-mediated immunity defect or for which the clinical course or management was complicated by HIV infection. Category C comprised AIDS-defining conditions.
  participants
    Asymptomatic or lymphadenopathy | 81 | 16 | 124 | 13 | 26 | 30 | 76 | 29 | 395
    Symptomatic, not AIDS | 17 | 1 | 48 | 23 | 21 | 24 | 23 | 18 | 175
    Acquired Immune Deficiency Syndrome (AIDS) | 21 | 1 | 49 | 18 | 26 | 24 | 5 | 39 | 183

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Event (AE): Interim Analysis
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. A list of all adverse events is reported in the "Other (Non-Serious) Adverse Events" section.
Time Frame: Baseline (Day 1) up to 31 January 2006 (up to Week 264)
Population: All participants receiving at least one dose of FPV or FPV/RTV in Study APV30005.
Measure: Number; unit: participants
Arm/Group | FPV Population (APV30001) | NFV Population (APV30001) | FPV Population (APV30002) | NFV Population (APV30002) | FPV/RTV QD Population (APV30003) | FPV/RTV BID Population (APV30003) | PI-Naïve Population (Other Studies) | PI-Experienced Population (Other Studies)
Number analyzed (Participants) | 119 | 18 | 221 | 54 | 73 | 78 | 104 | 86
participants | 117 | 16 | 215 | 52 | 72 | 75 | 95 | 68

2. Primary Outcome: Number of Participants With Any Adverse Event (AE): Final Analysis
Description: as for outcome 1
Time Frame: Post January 2006; for up to 241 weeks
Population: All participants who remained in the study after January 31, 2006.
Measure: Number; unit: participants
Arm/Group | Final Analysis Population (APV30005)
Number analyzed (Participants) | 111
participants | 95

3. Primary Outcome: Change From Baseline in the Indicated Clinical Chemistry Parameters at Weeks 48, 96, 120, 132, 168, 180, 204, and 216
Description: Fasting blood samples of participants were collected for the assessment of triglycerides (Tri.), cholesterol (Chol.), high density cholesterol (HDL), low density cholesterol (LDL), and fasting blood glucose (FBG). Change from Baseline at Weeks (W) 48, 96, 120, 132, 168, 180, 204, and 216 was calculated as the value at that particular week minus the value at Baseline (Day 1).
Time Frame: Baseline (Day 1) and Weeks 48, 96, 120, 132, 168, 180, 204, and 216
Population: All participants receiving at least one dose of FPV or FPV/RTV in Study APV30005. Only those participants contributing data at the indicated time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: milligrams per deciliter (mg/dl)
Arm/Group | FPV Population (APV30001) | NFV Population (APV30001) | FPV Population (APV30002) | NFV Population (APV30002) | FPV/RTV QD Population (APV30003) | FPV/RTV BID Population (APV30003) | PI-Naïve Population (Other Studies) | PI-Experienced Population (Other Studies)
Number analyzed (Participants) | 92 | 14 | 159 | 38 | 61 | 65 | 77 | 59
milligrams per deciliter (mg/dl)
  Tri.; W 48, n=54, 14, 159, 38, 61, 65, 77, 59 | 10 [-34 to 42] | -41 [-63 to -20] | 51 [14 to 118] | 20 [-19 to 57] | 9 [-25 to 44] | 14 [-69 to 66] | 5 [-27 to 58] | -54 [-96 to -12]
  Tri.; W 96, n=92, 13, 132 36, 47, 52, 67, 44 | 9 [-26 to 43] | -48 [-101 to 8] | 47 [10 to 101] | 15 [-22 to 48] | 16 [-51 to 40] | 34 [-21 to 118] | -5 [-35 to 42] | 7 [-3 to 41]
  Tri.; W 120, n=84, 14, 137, 33, 45, 49, 61, 40 | 15 [-24 to 59] | -33 [-77 to 0] | 43 [2 to 121] | -4 [-24 to 69] | 13 [-27 to 49] | 22 [-39 to 96] | -4 [-50 to 50] | -73 [-283 to 2]
  Tri.; W 132, n=82, 12, 128, 32, 40, 44, 61, 40 | 2 [-27 to 46] | -2 [-66 to 6] | 47 [-0 to 101] | 18 [-21 to 58] | 14 [-63 to 65] | 18 [-61 to 63] | 6 [-48 to 32] | -129 [-343 to 75]
  Tri.; W 168, n=71, 14, 123, 31, 31, 40, 20, 33 | 3 [-27 to 66] | -12 [-58 to 25] | 27 [-19 to 86] | 4 [-16 to 49] | 29 [-55 to 59] | 42 [-25 to 177] | 5 [-32 to 27] | -167 [-238 to -10]
  Tri.; W 180, n=73, 12, 114, 30, 33, 38, 61, 40 | 8 [-38 to 43] | -41 [-89 to 7] | 37 [4 to 87] | 18 [-16 to 81] | 13 [-27 to 63] | 8 [-95 to 112] | -2 [-38 to 20] | -170 [-267 to -56]
  Tri.; W 204, n=73, 12, 113, 23, 20, 26, 61, 40 | 2 [-26 to 44] | -36 [-88 to -14] | 43 [8 to 87] | 12 [-18 to 54] | 4 [-45 to 28] | 49 [-26 to 161] | 12 [-4 to 33] | NA [NA to NA] — No participants were analyzed in this arm at this time point.
  Tri.; W 216, n=76, 0, 111, 2, 5, 11, 61, 40 | 7 [-35 to 49] | NA [NA to NA] — No participants were analyzed in this arm at this time point. | 39 [4 to 97] | 98 [34 to 163] | -7 [-165 to 57] | 66 [-33 to 160] | NA [NA to NA] — No participants were analyzed in this arm at this time point. | NA [NA to NA] — No participants were analyzed in this arm at this time point.
  Chol.; W 48, n=54, 14, 159, 38, 61, 65, 77, 59 | 52 [23 to 70] | 3 [-32 to 13] | 53 [26 to 77] | 10 [-6 to 26] | 14 [-9 to 34] | 13 [-12 to 33] | 8 [-13 to 22] | 22 [-14 to 44]
  Chol.; W 96, n=92, 13, 132, 36, 47, 52, 67, 44 | 39 [19 to 58] | -3 [-16 to 25] | 46 [21 to 68] | 8 [-14 to 23] | 12 [-15 to 26] | 10 [-13 to 38] | 13 [-9 to 32] | 19 [1 to 57]
  Chol.; W 120, n=84, 14, 137, 33, 45, 49, 61, 40 | 42 [22 to 64] | -9 [-17 to 9] | 50 [23 to 73] | 9 [-15 to 23] | 11 [-16 to 25] | 22 [-8 to 31] | 13 [-10 to 30] | 32 [12 to 44]
  Chol.; W 132, n=82, 13, 128, 32, 40, 44, 61, 40 | 43 [22 to 72] | 14 [-23 to 32] | 47 [18 to 82] | 13 [-10 to 38] | 14 [-13 to 30] | -4 [-24 to 30] | 2 [-12 to 27] | 12 [-38 to 41]
  Chol.; W 168, n=71, 14, 123, 31, 31, 40, 20, 33 | 56 [28 to 78] | 6 [-18 to 38] | 47 [18 to 76] | 21 [-4 to 60] | 18 [-15 to 34] | 9 [-22 to 31] | 6 [-1 to 23] | 28 [19 to 52]
  Chol.; W 180, n=73, 12, 114, 30, 33, 38, 61, 40 | 54 [22 to 73] | -4 [-16 to 28] | 53 [24 to 78] | 19 [-4 to 40] | 3 [-8 to 34] | 9 [-19 to 27] | 5 [-1 to 17] | 43 [1 to 61]
  Chol.; W 204, n=73, 12, 113, 23, 20, 26, 61, 40 | 52 [18 to 76] | 5 [-32 to 22] | 53 [22 to 80] | 22 [-18 to 61] | -3 [-38 to 18] | 11 [-9 to 36] | -5 [-12 to 14] | NA [NA to NA] — No participants were analyzed in this arm at this time point.
  Chol.; W 216, n=76, 0, 111, 2, 5, 11, 61, 40 | 52 [25 to 79] | NA [NA to NA] — No participants were analyzed in this arm at this time point. | 47 [24 to 70] | 30 [24 to 35] | -65 [-82 to -48] | 28 [-8 to 34] | NA [NA to NA] — No participants were analyzed in this arm at this time point. | NA [NA to NA] — No participants were analyzed in this arm at this time point.
  HDL Chol.; W 48, n=54, 14, 159, 38, 61, 65, 77 59, | 10 [4 to 18] | -0.2 [-5 to 5] | 8 [2 to 15] | 3 [-5 to 8] | 6 [-1 to 10] | 2 [-4 to 11] | 3 [-3 to 8] | 8 [5 to 13]
  HDL Chol.; W 96, n=92, 13, 132, 36, 47, 52, 67, 44 | 12 [4 to 18] | 8 [1 to 16] | 12 [4 to 19] | 4 [-2 to 10] | 6 [-1 to 12] | 2 [-6 to 10] | 4 [-3 to 8] | 5 [4 to 13]
  HDL Chol.; W 120, n=84, 14, 137, 33, 45, 49, 61,40 | 12 [6 to 17] | 5 [1 to 11] | 12 [3 to 20] | 7 [0 to 15] | 8 [1 to 13] | 4 [-2 to 9] | 5 [-6 to 11] | 10 [9 to 20]
  HDL Chol.; W 132, n=82, 13, 128, 32, 40, 44, 61,40 | 13 [4 to 21] | 6 [-1 to 13] | 12 [7 to 20] | 9 [3 to 17] | 6 [3 to 15] | 5 [-2 to 12] | 3 [-6 to 11] | 16 [12 to 22]
  HDL Chol.; W 168, n=71, 14, 123, 31, 31, 40, 0, 0 | 17 [9 to 24] | 13 [3 to 21] | 17 [6 to 24] | 12 [3 to 17] | 8 [-1 to 15] | 2 [-5 to 8] | 10 [3 to 14] | 5 [4 to 24]
  HDL Chol.; W 180, n=73, 12, 114, 30, 33, 38, 61,40 | 17 [9 to 24] | 4 [1 to 16] | 15 [7 to 25] | 10 [3 to 17] | 7 [1 to 12] | 4 [-4 to 9] | 12 [NA to NA] — Only one participant was analyzed in this arm at this time point. | 18 [15 to 26]
  HDL Chol.; W 204, n=73, 10, 113, 23, 20, 26, 61,40 | 16 [8 to 26] | 10 [-0.2 to 16] | 17 [10 to 26] | 15 [2 to 22] | 6 [-0.19 to 15] | 2 [-7 to 12] | 3 [NA to NA] — Only one participant was analyzed in this arm at this time point. | NA [NA to NA] — No participants were analyzed in this arm at this time point.
  HDL Chol.; W 216, n=76, 0, 111, 2, 5, 11, 61, 40 | 16 [9 to 26] | NA [NA to NA] — No participants were analyzed in this arm at this time point. | 17 [7 to 25] | 4 [3 to 6] | 3 [-5 to 4] | 6 [-3 to 12] | NA [NA to NA] — No participants were analyzed in this arm at this time point. | NA [NA to NA] — No participants were analyzed in this arm at this time point.
  LDL Chol.; W 48, n=50, 13, 145, 35, 53, 50, 67, 48 | 32 [20 to 53] | 10 [-11 to 16] | 30 [10 to 53] | 0 [-8 to 19] | 2 [-24 to 21] | -1 [-15 to 24] | 3 [-13 to 21] | 17 [10 to 29]
  LDL Chol.; W 96, n=87, 12, 121, 34, 43, 43, 63, 37 | 25 [9 to 40] | -2 [-10 to 12] | 21 [4 to 45] | 1 [-20 to 17] | 3 [-20 to 15] | 0 [-18 to 27] | 7 [-12 to 25] | 15 [13 to 45]
  LDL Chol.; W 120, n=78, 13, 120, 29, 40, 39, 61,40 | 27 [10 to 44] | -4 [-11 to 8] | 21 [3 to 41] | -2 [-21 to 11] | -6 [-20 to 8] | 12 [-19 to 25] | 3 [-9 to 22] | 38 [22 to 61]
  LDL Chol.; W 132, n=78, 12, 117, 29, 36, 37, 58,34 | 25 [10 to 42] | 11 [-20 to 18] | 24 [-3 to 43] | 4 [-25 to 19] | -4 [-27 to 20] | -2 [-20 to 17] | 0 [-22 to 20] | 14 [14 to 15]
  LDL Chol.; W 168, n=63, 13, 115, 30, 28, 34, 0, 0 | 37 [13 to 54] | -5 [-17 to 20] | 18 [0.3 to 43] | 5 [-17 to 23] | -3 [-25 to 11] | -6 [-27 to 22] | -1 [-8 to 2] | 48 [24 to 72]
  LDL Chol.; W 180, n=67, 11, 111, 27, 29, 30, 61,40 | 27 [13 to 56] | 1 [-8 to 18] | 23 [4 to 49] | 2 [-18 to 14] | -2 [-16 to 17] | 4 [-20 to 18] | -7 [NA to NA] — Only one participant was analyzed in this arm at this time point. | 54 [48 to 60]
  LDL Chol.; W 204, n=70, 11, 105, 22, 19, 19, 61,40 | 35 [8 to 51] | 5 [-24 to 19] | 22 [2 to 46] | 13 [-18 to 40] | -14 [-32 to 12] | 1 [-26 to 25] | -45 [NA to NA] — Only one participant was analyzed in this arm at this time point. | NA [NA to NA] — No participants were analyzed in this arm at this time point.
  LDL Chol.; W 216, n=69, 0, 105, 2, 4, 10, 61, 40 | 33 [7 to 55] | NA [NA to NA] — No participants were analyzed in this arm at this time point. | 21 [-3 to 45] | 5 [-15 to 26] | -39 [-66 to -23] | 3 [-42 to 45] | NA [NA to NA] — No participants were analyzed in this arm at this time point. | NA [NA to NA] — No participants were analyzed in this arm at this time point.
  FBG; W 48, n=54, 14, 158, 36, 61, 65, 77, 59 | 7 [0 to 16] | -2 [-4 to 2] | 3.6 [-5 to 11] | -4 [-9 to 6] | 2 [-4 to 11] | 7 [-2 to 13] | 0 [-9 to 11] | 0 [-16 to 7]
  FBG; W 96, n=92, 13, 132, 34, 47, 52, 67, 44 | 4 [-4 to 11] | 0 [-5 to 4] | 1.8 [-4 to 11] | -5 [-11 to 0] | 0 [-9 to 9] | 4 [-5 to 14] | 0 [-11 to 7] | -5 [-11 to 5]
  FBG; W 120, n=84, 14, 136, 31, 44, 48, 61, 40 | 5 [-2 to 14] | -2 [-7 to 2] | 1.8 [-5 to 11] | -9 [-16 to -4] | 1 [-6 to 7] | 2 [-10 to 12] | 0 [-7 to 11] | -2 [-11 to 2]
  FBG; W 132, n=82, 13, 128, 30, 40, 44, 61, 40 | 0 [-5 to 13] | 0 [-5 to 2] | 0 [-7 to 11] | -4 [-5 to 4] | 0 [-9 to 5] | 0 [-10 to 7] | 7 [-2 to 16] | -14 [-21 to -8]
  FBG; W 168, n=71, 14, 123, 29, 31, 40, 0, 0 | 4 [-5 to 11] | 1 [-4 to 4] | 0 [-9 to 9] | -2 [-7 to 5] | 2 [-4 to 7] | -3 [-14 to 9] | 21 [13 to 24] | 0 [-2 to 2]
  FBG; W 180, n=73, 12, 112, 28, 33, 37, 61, 40 | 2 [-7 to 11] | -0.9 [-4 to 1] | 2.7 [-5 to 9.0] | -1.8 [-7 to 7] | 2 [-4 to 11] | 2 [-6 to 7] | 20 [14 to 29] | -1 [-5 to 3]
  FBG; W 204, n=73, 12, 115, 23, 20, 26, 61, 40 | 2 [-5 to 9] | 4 [-8 to 9] | 1.8 [-5 to 11] | 0 [-5 to 5] | 0 [-7 to 7] | 5 [-5 to 16] | 21 [14 to 25] | NA [NA to NA] — No participants were analyzed in this arm at this time point.
  FBG; W 216, n=75, 0, 110, 2, 5, 11, 61, 40 | 0 [-5 to 7] | NA [NA to NA] — No participants were analyzed in this arm at this time point. | 5.4 [-2 to 13] | 2 [-2 to 5] | 0 [-7 to 16] | 11 [-2 to 20] | NA [NA to NA] — No participants were analyzed in this arm at this time point. | NA [NA to NA] — No participants were analyzed in this arm at this time point.

4. Primary Outcome: Median Values of the Indicated Clinical Chemistry Parameters at Weeks 120, 180, 204, 216, and 432
Description: Fasting blood samples of participants were collected for the assessment of triglycerides, cholesterol, high density cholesterol (HDL), low density cholesterol (LDL), and fasting blood glucose (FBG).
Time Frame: Weeks 120, 180, 204, 216, and 432
Population: All participants who remained in the study after January 31, 2006. Only those participants contributing data at the indicated time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: milligrams per deciliter (mg/dl)
Arm/Group | Final Analysis Population (APV30005)
Number analyzed (Participants) | 106
milligrams per deciliter (mg/dl)
  Triglycerides; Week 120, n=14 | 237 [187 to 372]
  Triglycerides; Week 180, n=14 | 248 [193 to 312]
  Triglycerides; Week 204, n=106 | 137 [95 to 204]
  Triglycerides; Week 216, n=102 | 120 [92 to 192]
  Triglycerides; Week 432, n=40 | 132 [76 to 182]
  Cholesterol; Week 120, n=14 | 202 [183 to 284]
  Cholesterol; Week 180, n=14 | 206 [20 to 226]
  Cholesterol; Week 204, n=106 | 201 [166 to 232]
  Cholesterol; Week 216, n=102 | 205 [169 to 239]
  Cholesterol; Week 432, n=40 | 192 [168 to 233]
  HDL Cholesterol; Week 120, n=14 | 40 [34 to 45]
  HDL Cholesterol; Week 180, n=14 | 36 [34 to 47]
  HDL Cholesterol; Week 204, n=106 | 52 [42 to 61]
  HDL Cholesterol; Week 216, n=102 | 51 [44 to 62]
  HDL Cholesterol; Week 432, n=40 | 51 [44 to 57]
  LDL Cholesterol; Week 120, n=14 | 40 [34 to 45]
  LDL Cholesterol; Week 180, n=14 | 40 [34 to 48]
  LDL Cholesterol; Week 204, n=106 | 52 [42 to 61]
  LDL Cholesterol; Week 216, n=102 | 51 [44 to 62]
  LDL Cholesterol; Week 432, n=40 | 51 [44 to 57]
  FBG; Week 120, n=14 | 86 [79 to 97]
  FBG; Week 180, n=14 | 88 [85 to 92]
  FBG; Week 204, n=106 | 92 [81 to 97]
  FBG; Week 216, n=104 | 90 [81 to 97]
  FBG Cholesterol; Week 432, n=40 | 92 [83 to 100]

5. Primary Outcome: Change From Baseline in the Total Cholesterol/HDL Ratio at Weeks 48, 120, 180, 204, and 216
Description: blood samples of participants were collected for the assessment of the total cholesterol/HDL ratio. The ratio of total cholesterol/HDL was calculated by dividing the value of total cholesterol by the value of HDL. Change from Baseline at Weeks 48, 120, 180, 204, and 216 was calculated as the value at that particular week minus the value at Baseline (Day 1).
Time Frame: Baseline (Day 1) and Weeks 48, 120, 180, 204, and 216
Population: All participants receiving FPV or FPV/RTV in Study APV30005 having previously participated in Study APV30001 or Study APV30002. Only those participants contributing data at the indicated time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | FPV Population (APV30001) | NFV Population (APV30001) | FPV Population (APV30002) | NFV Population (APV30002)
Number analyzed (Participants) | 84 | 14 | 159 | 38
ratio
  Week 48, n=54, 14, 159, 38 | 0.1 [-0.4 to 0.8] | -0.4 [-1.0 to 0.6] | 0.4 [-0.3 to 1.2] | 0.1 [-0.3 to 0.5]
  Week 120, n=84, 14, 137, 33 | -0.2 [-0.7 to 0.4] | -0.6 [-1.1 to -0.2] | -0.1 [-0.8 to 0.7] | -0.2 [-0.7 to 0.1]
  Week 180, n=73, 12, 114, 30 | -0.4 [-1.1 to 0.2] | -0.6 [-1.6 to 0.1] | -0.3 [-1.0 to 0.4] | -0.3 [-1.3 to 0]
  Week 204, n=73, 12, 113, 23 | -0.3 [-1.0 to 0.1] | -0.6 [-1.7 to 0.1] | -0.4 [-1.0 to 0.1] | -0.4 [-0.9 to 0.23]
  Week 216, n=76, 0, 111, 2 | -0.5 [-1.0 to 0.2] | NA [NA to NA] — No participants were analyzed in this arm at this time point. | -0.5 [-1.1 to 0.1] | 0.3 [0.1 to 0.6]

6. Primary Outcome: Change From Baseline in the Total Cholesterol/HDL Ratio at Weeks 48, 96, 132, and 168
Description: Fasting blood samples of participants were collected for the assessment of the total cholesterol/HDL ratio. The ratio of total cholesterol/HDL was calculated by dividing the value of total cholesterol by the value of HDL. Change from Baseline at Weeks 48, 96, 132, and 168 was calculated as the value at that particular week minus the value at Baseline (Day 1).
Time Frame: Baseline (Day 1) and Weeks 48, 96, 132, and 168
Population: All participants receiving FPV or FPV/RTV in Study APV30005 having previously participated in Study APV30003 or other studies. Only those participants contributing data at the indicated time points were analyzed.
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | FPV/RTV QD Population (APV30003) | FPV/RTV BID Population (APV30003) | PI-Naïve Population (Other Studies) | PI-Experienced Population (Other Studies)
Number analyzed (Participants) | 61 | 65 | 45 | 7
ratio
  Week 48, n=61, 65 , 45, 7 | -0.4 [-1.1 to 0.4] | -0.3 [-1.1 to 0.8] | -0.1 [-0.8 to 0.8] | -0.8 [-0.8 to -0.1]
  Week 96, n=47, 52, 42, 5 | -0.5 [-1.4 to 0] | 0.1 [-0.8 to 0.8] | -0.1 [-0.7 to 0.4] | -0.3 [-0.5 to 0]
  Week 132, n=40, 44, 41, 4 | -0.4 [-1.5 to -0.1] | -0.6 [-1.6 to 0.5] | -0.2 [-1.1 to 1.0] | -1.5 [-2.7 to -0.3]
  Week 168, n=31, 40, 3, 5 | -0.3 [-1.4 to 0.3] | 0.2 [-1.0 to 0.5] | -0.6 [-1.0 to -0.4] | -1.4 [-1.4 to 0.1]

7. Primary Outcome: Median Value of the Total Cholesterol/HDL Ratio at Weeks 120, 180, 204, 216, and 432
Description: Fasting blood samples of participants were collected for the assessment of the total cholesterol/HDL ratio. The ratio of total cholesterol/HDL was calculated by dividing the value of total cholesterol by the value of HDL.
Time Frame: Weeks 120, 180, 204, 216, and 432
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Final Analysis Population (APV30005)
Number analyzed (Participants) | 106
ratio
  Week 120, n=14 | 5.5 [4.5 to 5.8]
  Week 180, n=14 | 5.5 [4.7 to 6.0]
  Week 204, n=106 | 3.7 [3.0 to 4.8]
  Week 216, n=102 | 3.5 [3.0 to 4.5]
  Week 432, n=40 | 4.0 [3.3 to 4.4]

8. Primary Outcome: Change From Baseline in Aspartate Aminotransferase (AST), Alanine Transaminase (ALT), and Serum Lipase at Weeks 48, 120, 180, 204, and 216
Description: Blood samples of participants were collected for the assessment of AST, ALT, and serum lipase. Change from Baseline at Weeks 48, 120, 180, 204, and 216 was calculated as the value at that particular week minus the value at Baseline (Day 1).
Time Frame: Baseline (Day 1) and Weeks 48, 120, 180, 204, and 216
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: units per liter (U/L)
Arm/Group | FPV Population (APV30001) | NFV Population (APV30001) | FPV Population (APV30002) | NFV Population (APV30002)
Number analyzed (Participants) | 118 | 17 | 217 | 47
units per liter (U/L)
  AST; Week 48, n=117, 17, 215, 47 | -7 [-14 to -1] | -2 [-3 to 5] | -7 [-17 to -1] | 0 [-5 to 5]
  AST; Week 120, n=96, 15, 182, 40 | -8 [-19 to -1] | 0 [-8 to 4] | -8 [-19 to -2] | 1 [-3 to 4]
  AST; Week 180, n=80, 12, 154, 33 | -10 [-19 to -3] | 2 [-5 to 4] | -7 [-18 to -1] | -2 [-4 to 2]
  AST; Week 204, n=77, 12, 151, 27 | -7 [-18 to -1] | 3 [-4 to 6] | -7 [-18 to -1] | -2 [-4 to 2]
  AST; Week 216, n=79, 0, 142, 4 | -9 [-16 to -1] | NA [NA to NA] — No participants were analyzed in this arm at this time point. | -7 [-17 to 0] | 1 [-7 to 8]
  ALT; Week 48, n=117, 17, 216, 47 | -5 [-21 to 2] | 0 [-3 to 4] | -8 [-19 to 1] | 2 [-2 to 8]
  ALT; Week 120, n=96, 15, 182, 40 | -9 [-29 to 2] | -1 [-6 to 7] | -8 [-20 to 0] | 4 [-6 to 8]
  ALT; Week 180, n=81, 12, 155, 33 | -10 [-27 to -1] | 3 [-3 to 5] | -6 [-19 to 5] | 1 [-5 to 6]
  ALT; Week 204, n=77, 12, 152, 27 | -10 [-26 to 0] | 2 [-1 to 9] | -5 [-19 to 4] | -1 [-7 to 5]
  ALT; Week 216, n=79, 0, 142, 4 | -10 [-27 to 2] | NA [NA to NA] — No participants were analyzed in this arm at this time point. | -6 [-18 to 2] | -3 [-11 to 9]
  Serum lipase; Week 48, n=118, 17, 217, 47 | 4 [-2 to 10] | 1 [-8 to 5] | 0 [-7 to 7] | -2 [-6 to 1]
  Serum lipase; Week 120, n=95, 15, 184, 40 | 4 [-4 to 9] | 4 [-1 to 6] | -1 [-6 to 6] | 2 [-4 to 7]
  Serum lipase; Week 180, n=81, 12, 156, 33 | 4 [-3 to 9] | -0.5 [-6 to 4] | 1 [-5 to 6] | 1 [-5 to 3]
  Serum lipase;Week 204, n=78, 12, 153, 27 | 3 [-4 to 10] | 0 [-5 to 3] | 1 [-5 to 7] | 2 [-4 to 6]
  Serum lipase; Week 216, n=80, 0, 143, 4 | 5 [-2 to 11] | NA [NA to NA] — No participants were analyzed in this arm at this time point. | 0 [-6 to 9] | -3 [-27 to 5]

9. Primary Outcome: Change From Baseline in Aspartate Aminotransferase (AST), Alanine Transaminase (ALT), and Serum Lipase at Weeks 48, 96, 132, and 168
Description: Blood samples of participants were collected for the assessment of AST, ALT, and serum lipase. Change from Baseline at Weeks 48, 96, 132, and 168 was calculated as the value at that particular week minus the value at Baseline (Day 1).
Time Frame: Baseline (Day 1) and Weeks 48, 96, 132, and 168
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: units per liter (U/L)
Arm/Group | FPV/RTV QD Population (APV30003) | FPV/RTV BID Population (APV30003) | PI-Naïve Population (Other Studies) | PI-Experienced Population (Other Studies)
Number analyzed (Participants) | 73 | 78 | 83 | 65
units per liter (U/L)
  AST; Week 48, n=73, 78, 83, 65 | -6 [-14 to 3] | -5 [-15 to -1] | 1 [-3 to 4] | 0 [-6 to 6]
  AST; Week 96, n=57, 63, 73, 49 | -6 [-12 to 6] | -4 [-18 to 2] | 1 [-3 to 3] | -1 [-9 to 4]
  AST; Week 132, n=50, 57, 64, 46 | -6 [-13 to -1] | -4 [-14 to 2] | 2 [-3 to 5] | 1 [-5 to 8]
  AST; Week 168, n=45, 48, 20, 36 | -6 [-14 to 1] | -6 [-17 to -1] | 2 [-1 to 5] | -1 [-10 to 5]
  ALT; Week 48, n=70, 78, 83, 65 | -2 [-13 to 4] | -6 [-21 to 1] | 2 [-2 to 8] | 0 [-9 to 12]
  ALT; Week 96, n=59, 63, 73, 49 | -4 [-13 to 9] | -3 [-21 to 3] | 2 [-3 to 6] | 1 [-10 to 6]
  ALT; Week 132, n=51, 58, 64, 46 | -2 [-17 to 8] | -4 [-18 to 3] | 2 [-2 to 8] | 2 [-10 to 8]
  ALT; Week 168, n=45, 48, 20, 37 | -5 [-23 to 4] | -5 [-22 to 4] | 6 [-1 to 9] | -3 [-16 to 6]
  Serum lipase; Week 48, n=72, 78, 57, 64 | 1 [-5 to 8] | 2 [-4 to 9] | 1 [-3 to 7] | 1 [-4 to 6]
  Serum lipase; Week 96, n=59, 63, 52, 49 | 3 [-4 to 10] | 4 [-5 to 12] | 0 [-3 to 3] | 3 [-4 to 11]
  Serum lipase; Week 132, n=52, 58, 47, 46 | 2 [-4 to 10] | 4 [-1 to 13] | 1 [-3 to 5] | 2 [-4 to 11]
  Serum lipase; Week 168, n=45, 48, 7, 37 | 0 [-8 to 6] | 2 [-1 to 11] | -5 [-14 to 8] | 3 [-6 to 16]

10. Primary Outcome: Median Aspartate Aminotransferase (AST), Alanine Transaminase (ALT), and Serum Lipase Values at Weeks 120, 180, 204, 216, and 432
Description: Blood samples of participants were collected for the assessment of AST, ALT, and serum lipase.
Time Frame: Weeks 120, 180, 204, 216, and 432
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: units per liter (U/L)
Arm/Group | Final Analysis Population (APV30005)
Number analyzed (Participants) | 107
units per liter (U/L)
  AST; Week 120, n=14 | 18 [17 to 22]
  AST; Week 180, n=14 | 21 [19 to 23]
  AST; Week 204, n=107 | 20 [16 to 23]
  AST; Week 216, n=106 | 21 [18 to 25]
  AST; Week 432, n=41 | 21 [17 to 24]
  ALT; Week 120, n=14 | 18 [14 to 27]
  ALT; Week 180, n=14 | 32 [22 to 36]
  ALT; Week 204, n=107 | 19 [13 to 25]
  ALT; Week 216, n=106 | 19 [14 to 25]
  ALT; Week 432, n=41 | 19 [15 to 24]
  Serum lipase;Week 120, n=14 | 47 [31 to 53]
  Serum lipase; Week 180, n=14 | 39 [29 to 49]
  Serum lipase; Week 204, n=107 | 34 [27 to 44]
  Serum lipase; Week 216, n=106 | 36 [26 to 43]
  Serum lipase; Week 432, n=41 | 36 [30 to 47]

11. Secondary Outcome: Percentage of Participants With Plasma HIV-1 Ribonucleic Acid (RNA) <400 and <50 Copies Per Milliliter at Baseline and Weeks 48, 120, 180, and 216 (MD=F and Observed)
Description: Blood samples of participants were collected for the assessment of HIV-1RNA copies in plasma. Viral load, measured in RNA copies per milliliter of plasma, is an efficacy measure for antiretroviral drugs. In the MD=F analysis, participants who had missing data at or had discontinued the study prior to a certain time point are classified as non-responders. In the observed analysis (OA), data are presented for the number of participants still enrolled in the study at a certain time point. Participants in the NFV populations had received antiretroviral therapy prior to Baseline.
Time Frame: Baseline and Weeks 48, 120, 180, and 216
Population: All participants receiving FPV or FPV/RTV in Study APV30005 having previously participated in Study APV30001 or Study APV30002. No participants were analyzed in the NPV APV30001 arm due to their small number.
Measure: Number; unit: percentage of participants
Arm/Group | FPV Population (APV30001) | NFV Population (APV30001) | FPV Population (APV30002) | NFV Population (APV30002)
Number analyzed (Participants) | 119 | 0 | 221 | 54
percentage of participants
  Baseline <400 copies, n=119, 219, 54; MD=F | 1 |  | 0 | 61
  Week 48 <400 copies, n=119, 219, 54; MD=F | 92 |  | 94 | 85
  Week 120 <400 copies, n=119, 219, 54; MD=F | 76 |  | 77 | 69
  Week 180 <400 copies, n=119, 219, 54; MD=F | 66 |  | 68 | 54
  Week 216 <400 copies, n=119, 219, 0; MD=F | 62 |  | 61 | NA — No participants were analyzed in this arm at this time point.
  Baseline <400 copies, n=119, 219, 54; observed | 1 |  | 0 | 61
  Week 48 <400 copies, n=118, 216, 49; observed | 93 |  | 95 | 94
  Week 120 <400 copies, n=96, 181, 40; observed | 95 |  | 93 | 93
  Week 180 <400 copies, n=82, 158, 34; observed | 95 |  | 94 | 85
  Week 216 <400 copies, n=80, 142, 0; observed | 93 |  | 94 | NA — No participants were analyzed in this arm at this time point.
  Baseline <50 copies, n=119, 219, 54; MD=F | 1 |  | 0 | 46
  Week 48 <50 copies, n=119, 219, 54; MD=F | 80 |  | 76 | 59
  Week 120 <50 copies, n=119, 219, 54; MD=F | 71 |  | 66 | 61
  Week 180 <50 copies, n=119, 219, 54; MD=F | 61 |  | 63 | 48
  Week 216 <50 copies, n=119, 219, 0; MD=F | 58 |  | 58 | NA — No participants were analyzed in this arm at this time point.
  Baseline <50 copies, n=119, 219, 54; observed | 1 |  | 0 | 46
  Week 48 <50 copies, n=118, 216, 49; observed | 81 |  | 77 | 65
  Week 120 <50 copies, n=96, 181, 40; observed | 88 |  | 80 | 83
  Week 180 <50 copies, n=82, 158, 34; observed | 88 |  | 88 | 76
  Week 216 <50 copies, n=80, 142, 0; observed | 86 |  | 89 | NA — No participants were analyzed in this arm at this time point.

12. Secondary Outcome: Percentage of Participants With Plasma HIV-1RNA <400 and <50 Copies Per Milliliter at Baseline and Weeks 12, 24, 48, 60, 96, and 132 (MD=F and Observed)
Description: Blood samples of participants were collected for the assessment of HIV-1RNA copies in plasma. Viral load, measured in RNA copies per milliliter of plasma, is an efficacy measure for antiretroviral drugs. In the MD=F analysis, participants who had missing data at or had discontinued the study prior to a certain time point are classified as non-responders. In the observed analysis (OA), data are presented for the number of participants still enrolled in the study at a certain time point.
Time Frame: Baseline and Weeks 12, 24, 48, 60, 96, and 132
Population: All participants receiving FPV or FPV/RTV in Study APV3005 having participated in Study APV30003 or other studies. The PI-naïve and PI-experienced populations (other studies) had received antiretroviral therapy prior to Baseline.
Measure: Number; unit: percentage of participants
Arm/Group | FPV/RTV QD Population (APV30003) | FPV/RTV BID Population (APV30003) | PI-Naïve Population (Other Studies) | PI-Experienced Population (Other Studies)
Number analyzed (Participants) | 73 | 78 | 104 | 86
percentage of participants
  Baseline <400 copies, n=73, 78, 104, 86; MD=F | 0 | 1 | 84 | 59
  Week 12 <400 copies, n=73, 78, 104, 86; MD=F | 75 | 82 | 82 | 52
  Week 24 <400 copies, n=73, 78, 104, 86; MD=F | 79 | 79 | 85 | 60
  Week 48 <400 copies, n=73, 78, 104, 86; MD=F | 71 | 78 | 78 | 50
  Week 60 <400 copies, n=73, 78, 104, 86; MD=F | 70 | 77 | 74 | 51
  Week 96 <400 copies, n=73, 78, 104, 86; MD=F | 58 | 62 | 67 | 45
  Week 132 <400 copies, n=73, 78, 104, 86; MD=F | 49 | 60 | 60 | 41
  Baseline <400 copies, n=73, 78, 92, 82; observed | 0 | 1 | 95 | 62
  Week 12 <400 copies, n=69, 78, 92, 79; observed | 80 | 82 | 92 | 57
  Week 24 <400 copies, n=73, 75, 93, 79; observed | 79 | 83 | 95 | 66
  Week 48 <400 copies, n=73, 77, 85, 68; observed | 71 | 79 | 95 | 63
  Week 60 <400 copies, n=71, 76, 81, 58; observed | 72 | 79 | 95 | 76
  Week 96 <400 copies, n=60, 62, 75, 51; observed | 70 | 77 | 93 | 76
  Week 132 <400 copies,n=50, 58, 65, 46; observed | 72 | 81 | 95 | 76
  Baseline <50 copies, n=73, 78, 104, 86; MD=F | 0 | 0 | 59 | 44
  Week 12 <50 copies, n=73, 78, 104, 86; MD=F | 47 | 47 | 78 | 40
  Week 24 <50 copies, n=73, 78, 104, 86; MD=F | 63 | 64 | 78 | 42
  Week 48 <50 copies, n=73, 78, 104, 86; MD=F | 49 | 60 | 69 | 42
  Week 60 <50 copies, n=73, 78, 104, 86; MD=F | 51 | 59 | 68 | 41
  Week 96 <50 copies, n=73, 78, 104, 86; MD=F | 45 | 51 | 61 | 37
  Week 132 <50 copies, n=73, 78, 104, 86; MD=F | 37 | 45 | 53 | 40
  Baseline <50 copies, n=73, 78, 92, 82; observed | 0 | 0 | 66 | 46
  Week 12 <50 copies, n=69, 78, 92, 79; observed | 49 | 47 | 88 | 43
  Week 24 <50 copies, n=73, 75, 93, 79; observed | 63 | 67 | 87 | 46
  Week 48 <50 copies, n=73, 77, 85, 68; observed | 49 | 61 | 85 | 53
  Week 60 <50 copies, n=71, 76, 81, 58; observed | 52 | 61 | 88 | 60
  Week 96 <50 copies, n=60, 62, 75, 51; observed | 55 | 65 | 84 | 63
  Week 132 <50 copies, n=50, 58, 65, 46; observed | 54 | 60 | 85 | 74

13. Secondary Outcome: Percentage of Participants With Plasma HIV-1RNA <50 Copies Per Milliliter at Baseline and Weeks 120, 180, 240, 300, 360, 420, and 432 (Observed)
Description: Blood samples of participants were collected for the assessment of HIV-1RNA copies in plasma. Viral load, measured in RNA copies per milliliter of plasma,is an efficacy measure for antiretroviral drugs.
Time Frame: Baseline and Weeks 120, 180, 240, 300, 360, 420, and 432
Population: All participants who remained in the study after January 31, 2006. Only those participants contributing data at the indicated time points were analyzed. In the observed analysis, data are presented for the number of participants still enrolled in the study who are classified as responders.
Measure: Number; unit: percentage of participants
Arm/Group | Final Analysis Population (APV30005)
Number analyzed (Participants) | 101
percentage of participants
  Week 120 <50 copies, n=14; observed | 93
  Week 180 <50 copies, n=14; observed | 86
  Week 240 <50 copies, n=101; observed | 87
  Week 300 <50 copies, n=82; observed | 93
  Week 360 <50 copies, n=53; observed | 89
  Week 420 <50 copies, n=52; observed | 92
  Week 432 <50 copies, n=41; observed | 93

14. Secondary Outcome: Cluster of Differentiation Antigen 4 (CD4+) Cell Count at Baseline and Weeks 48, 120, 168, 180, 204, and 216: Observed Analysis
Description: Blood samples of participants were collected for the assessment of CD4+ cell count. CD4+ cells are white blood cells that are important in fighting infection. HIV infects CD4+ cells, replicates in them, and destroys them. CD4+ cell count provides a measure of the status of the immune system and to what extent it is affected by HIV.
Time Frame: Baseline and Weeks 48, 120, 168, 180, 204, and 216
Population: All participants receiving FPV or FPV/RTV in Study APV30005 having previously participated in Study APV30001 or Study APV30002. Only those participants contributing data at the indicated time points were analyzed. Participants in the NFV populations had received antiretroviral therapy prior to Baseline.
Measure: Median (Full Range); unit: cells per millimeters cubed (cells/mm^3)
Arm/Group | FPV Population (APV30001) | NFV Population (APV30001) | FPV Population (APV30002) | NFV Population (APV30002)
Number analyzed (Participants) | 119 | 18 | 219 | 52
cells per millimeters cubed (cells/mm^3)
  Baseline, n=119, 18, 219, 52 | 211 [2 to 1136] | 505 [179 to 1788] | 167 [1 to 813] | 297 [5 to 755]
  Week 48, n=117, 17, 211, 49 | 426 [40 to 1326] | 499 [179 to 1367] | 396 [58 to 1188] | 377 [13 to 884]
  Week 120, n=95, 15, 177, 40 | 512 [116 to 1289] | 613 [274 to 1406] | 475 [90 to 1595] | 439 [124 to 888]
  Week 168, n=81, 12, 160, 37 | 594 [147 to 1534] | 608 [287 to 1069] | 506 [67 to 1299] | 422 [83 to 835]
  Week 180, n=78, 9, 153, 33 | 541 [418 to 765] | 447 [180 to 768] | 494 [113 to 1261] | 413 [129 to 970]
  Week 204, n=75, 11, 145, 27 | 535 [377 to 709] | 563 [226 to 998] | 494 [110 to 1420] | 459 [115 to 911]
  Week 216, n=77, 0, 138, 4 | 608 [477 to 846] | NA [NA to NA] — No participants were analyzed in this arm at this time point. | 534 [117 to 1687] | 548 [102 to 641]

15. Secondary Outcome: Cluster of Differentiation Antigen 4 (CD4+) Cell Count at Baseline and Weeks 24, 48, 96, 132, and 168: Observed Analysis
Description: as for outcome 14
Time Frame: Baseline and Weeks 24, 48, 96, 132, and 168
Population: All participants receiving FPV or FPV/RTV in Study APV30005 having previously participated in Study APV30003 and other studies. Only those participants contributing data at the indicated time points were analyzed. The PI-naїve and PI-experienced populations (other studies) had received antiretroviral therapy prior to Baseline.
Measure: Median (Full Range); unit: cells per millimeters cubed (cells/mm^3)
Groups:
- PI-Naïve Population (Other Studies): FFPV +/- RTV + background regimen in participants who were PI-naïve prior to enrollment in the parent study
Arm/Group | FPV/RTV QD Population (APV30003) | FPV/RTV BID Population (APV30003) | PI-Naïve Population (Other Studies) | PI-Experienced Population (Other Studies)
Number analyzed (Participants) | 73 | 78 | 94 | 76
cells per millimeters cubed (cells/mm^3)
  Baseline, n=72, 78, 94, 76 | 311 [6 to 1171] | 304 [41 to 845] | 477 [130 to 1224] | 361 [6 to 1354]
  Week 24, n=71, 73, 92, 75 | 367 [69 to 1391] | 348 [101 to 1051] | 520 [128 to 1266] | 399 [28 to 1120]
  Week 48, n=73, 77, 85, 68 | 374 [66 to 914] | 386 [99 to 965] | 582 [42 to 1194] | 418 [10 to 1121]
  Week 96, n=58, 62, 73, 50 | 409 [179 to 868] | 417 [82 to 744] | 567 [82 to 1342] | 463 [21 to 929]
  Week 132, n=50, 56, 64, 47 | 395 [120 to 1015] | 386 [38 to 820] | 642 [159 to 1193] | 486 [16 to 1769]
  Week 168, n=40, 47, 20, 39 | 513 [133 to 1069] | 409 [59 to 1097] | 619 [260 to 1312] | 460 [51 to 890]

16. Secondary Outcome: Median Plasma HIV-1 RNA at Baseline and Weeks 24, 48, 72, 96, 120, 144, 168, 180, 204, and 216
Description: Blood samples of participants were collected for the assessment of plasma HIV-1 RNA.
Time Frame: Baseline and Weeks 24, 48, 72, 96, 120, 144, 168, 180, 204, and 216
Population: All participants receiving FPV or FPV/RTV in Study APV30005 having previously particpated in Study APV30001 or Study APV30002. Only those participants contributing data at the indicated time points were analyzed. Participants in the NFV populations had received antiretroviral therapy prior to Baseline.
Measure: Median (Full Range); unit: log 10 copies per milliliter
Arm/Group | FPV Population (APV30001) | NFV Population (APV30001) | FPV Population (APV30002) | NFV Population (APV30002)
Number analyzed (Participants) | 119 | 18 | 221 | 54
log 10 copies per milliliter
  Baseline, n=119, 18, 221, 54 | 4.82 [1.69 to 7.4] | 1.69 [1.69 to 5.6] | 4.82 [2.65 to 7.29] | 1.78 [1.69 to 5.66]
  Week 24, n=119, 17, 217, 51 | 1.69 [1.69 to 5.8] | 1.69 [1.69 to 5.7] | 1.69 [1.69 to 5.49] | 1.69 [1.69 to 5.34]
  Week 48, n=118, 17, 218, 49 | 1.69 [1.69 to 5.9] | 1.69 [1.69 to 5.4] | 1.69 [1.69 to 5.03] | 1.69 [1.69 to 4.13]
  Week 72, n=113, 15, 204, 46 | 1.69 [1.69 to 4.8] | 1.69 [1.69 to 3.5] | 1.69 [1.69 to 5.83] | 1.69 [1.69 to 5.34]
  Week 96, n=106, 15, 192, 43 | 1.69 [1.69 to 4.7] | 1.69 [1.69 to 3.6] | 1.69 [1.69 to 5.38] | 1.69 [1.69 to 1.69]
  Week 120, n=96, 15, 183, 40 | 1.69 [1.69 to 4.9] | 1.69 [1.69 to 3.1] | 1.69 [1.69 to 5.53] | 1.69 [1.69 to 3.60]
  Week 144, n=89, 15, 173, 39 | 1.69 [1.69 to 4.2] | 1.69 [1.69 to 3.9] | 1.69 [1.69 to 5.38] | 1.69 [1.69 to 3.82]
  Week 168, n=81, 14, 160, 38 | 1.69 [1.69 to 4.8] | 1.69 [1.69 to 4.0] | 1.69 [1.69 to 5.44] | 1.69 [1.69 to 4.27]
  Week 180, n=82, 12, 159, 34 | 1.69 [1.69 to 4.7] | 1.69 [1.69 to 3.3] | 1.69 [1.69 to 4.71] | 1.69 [1.69 to 3.95]
  Week 204, n=78, 12, 153, 27 | 1.69 [1.69 to 3.8] | 1.69 [1.69 to 3.5] | 1.69 [1.69 to 5.26] | 1.69 [1.69 to 2.91]
  Week 216, n=80, 0, 143, 4 | 1.69 [1.69 to 5.4] | NA [NA to NA] — No participants were analyzed in this arm at this time point. | 1.69 [1.69 to 5.59] | 1.69 [1.69 to 1.69]

17. Secondary Outcome: Median Plasma HIV-1 RNA at Baseline and Weeks 12, 24, 48, 72, 96, 132, and 168
Description: Blood samples of participants were collected for the assessment of plasma HIV-1 RNA.
Time Frame: Baseline and Weeks 12, 24, 48, 72, 96, 132, and 168
Population: All participants receiving FPV or FPV/RTV in Study APV30005 having previously participated in Study APV30003 or other studies. Only those participants contributing data at the indicated time points were analyzed. The PI naïve and PI-experienced populations (other studies) had received antiretroviral therapy prior to Baseline.
Measure: Median (Full Range); unit: log 10 copies per milliliter
Arm/Group | FPV/RTV QD Population (APV30003) | FPV/RTV BID Population (APV30003) | PI-Naïve Population (Other Studies) | PI-Experienced Population (Other Studies)
Number analyzed (Participants) | 73 | 78 | 93 | 82
log 10 copies per milliliter
  Baseline, n=73, 78, 92, 82 | 3.96 [3.0 to 5.8] | 4.06 [2.3 to 5.9] | 1.7 [1.7 to 4.9] | 1.81 [1.7 to 6.2]
  Week 12, n=69, 78, 92, 79 | 1.7 [1.7 to 5.3] | 1.81 [1.7 to 5.8] | 1.7 [1.7 to 6.0] | 2.03 [1.7 to 5.9]
  Week 24, n=73, 75, 93, 79 | 1.69 [1.69 to 4.8] | 1.69 [1.69 to 5.6] | 1.7 [1.7 to 5.5] | 1.9 [1.7 to 5.7]
  Week 48, n=73, 77, 85, 68 | 1.71 [1.7 to 4.5] | 1.69 [1.69 to 5.8] | 1.7 [1.7 to 5.3] | 1.7 [1.7 to 5.1]
  Week 72, n=65, 73, 80, 53 | 1.72 [1.7 to 5.5] | 1.69 [1.69 to 5.4] | 1.7 [1.7 to 4.7] | 1.7 [1.7 to 5.3]
  Week 96, n=60, 62, 75, 51 | 1.69 [1.69 to 4.9] | 1.69 [1.69 to 5.2] | 1.7 [1.7 to 5.4] | 1.7 [1.7 to 5.8]
  Week 132, n=50, 58, 65, 46 | 1.69 [1.69 to 4.8] | 1.69 [1.69 to 5.8] | 1.7 [1.7 to 4.0] | 1.7 [1.7 to 5.3]
  Week 168, n=44, 48, 20, 39 | 1.69 [1.69 to 4.8] | 1.69 [1.69 to 4.9] | 1.7 [1.7 to 2.8] | 1.7 [1.7 to 4.5]

18. Secondary Outcome: Median Plasma HIV-1 RNA at Weeks 180, 240, 300, 360, 420, and 432
Description: Blood samples of participants were collected for the assessment of plasma HIV-1 RNA.
Time Frame: Weeks 180, 240, 300, 360, 420, and 432
Population: as for outcome 4
Measure: Median (Full Range); unit: log 10 copies per milliliters
Arm/Group | Final Analysis Population (APV30005)
Number analyzed (Participants) | 101
log 10 copies per milliliters
  Week 180, n=14 | 1.7 [1.7 to 4.1]
  Week 240, n=101 | 1.7 [1.7 to 4.4]
  Week 300, n=82 | 1.7 [1.7 to 4.5]
  Week 360, n=53 | 1.7 [1.7 to 4.6]
  Week 420, n=52 | 1.7 [1.7 to 4.9]
  Week 432, n=41 | 1.7 [1.7 to 4.7]

19. Secondary Outcome: Number of Participants With HIV-1 Disease Progression to CDC Class C, or New CDC Class C or Death, From Baseline
Description: The number of participants with progression of HIV-1 disease were assessed using the CDC classification of HIV-1: class A, asymptomatic or lymphadenopathy; class B: symptomatic, but not AIDS; class C, AIDS. A participant is considered to have had a disease progression if they report a CDC Class C event for the first time, if they report a new CDC Class C event, or if they experience any fatal adverse event during the study.
Time Frame: Baseline (Day 1) up to 31 January 2006 (up to Week 264)
Population: All participants receiving at least one dose of FPV or FPV/RTV in Study APV30005.
Measure: Number; unit: participants
Arm/Group | FPV Population (APV30001) | NFV Population (APV30001) | FPV Population (APV30002) | NFV Population (APV30002) | FPV/RTV QD Population (APV30003) | FPV/RTV BID Population (APV30003) | PI-Naïve Population (Other Studies) | PI-Experienced Population (Other Studies)
Number analyzed (Participants) | 119 | 18 | 221 | 54 | 73 | 78 | 104 | 86
participants
  CDC class A to CDC class C | 0 | 0 | 3 | 0 | 0 | 1 | 0 | 0
  CDC class B to CDC class C | 3 | 0 | 5 | 3 | 1 | 0 | 0 | 1
  CDC class C to new CDC class C | 1 | 0 | 2 | 2 | 0 | 0 | 0 | 1
  CDC class A, B, or C to death (on treatment) | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0

20. Secondary Outcome: Number of Participants Enrolled in Studies APV30001 and APV300002 With the Indicated HIV-associated Conditions
Description: The number of participants with the indicated HIV-associated conditions were assessed, excluding recurrences.
Time Frame: Baseline (Day 1) up to 31 January 2006 (up to Week 264)
Population: All participants receiving FPV or NFV in Studies APV30001 and APV30002.
Measure: Number; unit: participants
Arm/Group | FPV Population (APV30001) | NFV Population (APV30001) | FPV Population (APV30002) | NFV Population (APV30002)
Number analyzed (Participants) | 119 | 18 | 221 | 54
participants
  Candidiasis, oropharyngeal | 4 | 0 | 7 | 0
  Herpes zoster | 0 | 0 | 3 | 3
  Diarrhea lasting >1 month | 1 | 0 | 1 | 2
  Candidiasis, vulvovaginal | 1 | 0 | 0 | 0
  Cervical dysplasia | 1 | 0 | 0 | 0
  Fever lasting >1 month | 1 | 0 | 0 | 0
  Hairy leukoplakia, oral | 1 | 0 | 1 | 0
  Peripheral neuropathy | 1 | 0 | 2 | 0
  Cytomegalovirus retinitis | 1 | 0 | 0 | 0
  Herpes simplex | 1 | 0 | 1 | 0
  Mycobacterium tuberculosis, any site | 0 | 0 | 2 | 1
  Encepathopathy, HIV-related | 0 | 0 | 1 | 0
  Kaposis's sarcoma, cutaneous | 0 | 0 | 1 | 0
  Lymphoma,immunoblastic | 0 | 0 | 1 | 0
  Mycobacterium avium complex/ M kansaii | 0 | 0 | 1 | 0
  Pneumocystis carinii pneumonia | 0 | 0 | 1 | 0
  Progressive multifocal leukoencephalopathy | 0 | 0 | 1 | 0
  Toxoplasmosis of brain | 1 | 0 | 0 | 0
  Non-CDC HIV-associated conditions | 0 | 0 | 8 | 0

21. Secondary Outcome: Number of Participants Enrolled in Study APV30003 and Other Studies With the Indicated HIV-associated Conditions
Description: The number of participants with the indicated HIV-associated conditions were assessed.
Time Frame: Baseline (Day 1) up to 31 January 2006 (up to Week 264)
Population: All participants receiving FPV/RTV in Study APV30005 having previously participated in Study APV30003 or other studies.
Measure: Number; unit: participants
Arm/Group | FPV/RTV QD Population (APV30003) | FPV/RTV BID Population (APV30003) | PI-Naïve Population (Other Studies) | PI-Experienced Population (Other Studies)
Number analyzed (Participants) | 73 | 78 | 104 | 86
participants
  Candidiasis, oropharyngeal | 5 | 0 | 0 | 0
  Hairy leukoplakia, oral | 1 | 0 | 0 | 1
  Peripheral neuropathy | 1 | 1 | 0 | 0
  Diarrhea lasting >1 month | 0 | 1 | 0 | 0
  Herpes Zoster | 1 | 0 | 1 | 0
  Mycobacterium tuberculosis, any site | 1 | 0 | 0 | 0
  Other, Non-CDC HIV associated condition | 1 | 0 | 1 | 0

ADVERSE EVENTS:
Arm/Group | FPV Population (APV30001) | NFV Population (APV30001) | FPV Population (APV30002) | NFV Population (APV30002) | FPV/RTV QD Population (APV30003) | FPV/RTV BID Population (APV30003) | PI-Naïve Population (Other Studies) | PI-Experienced Population (Other Studies) | Final Analysis Population (APV30005)
Serious Adverse Events (participants affected / at risk) | 33/119 | 1/18 | 62/221 | 7/54 | 20/73 | 14/78 | 7/104 | 13/86 | 15/111
Other Adverse Events (participants affected / at risk) | 115/119 | 16/18 | 209/221 | 53/54 | 68/73 | 73/78 | 76/104 | 40/86 | 82/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | FPV Population (APV30001) (N=119) | NFV Population (APV30001) (N=18) | FPV Population (APV30002) (N=221) | NFV Population (APV30002) (N=54) | FPV/RTV QD Population (APV30003) (N=73) | FPV/RTV BID Population (APV30003) (N=78) | PI-Naïve Population (Other Studies) (N=104) | PI-Experienced Population (Other Studies) (N=86) | Final Analysis Population (APV30005) (N=111)
Anogenital warts (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis of male external genital organ (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastroenteritis salmonella (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Orchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 3 | 0 | 2 | 0 | 0 | 0 | 0
Scrotal abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Syphilis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lobar pneumonia (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1
Osteomyelitis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Bronchopneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Localised infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Meningitis viral (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia primary atypical (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Superinfection lung (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Abscess limb (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Meningitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hepatitis C (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Leishmaniasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Perianal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Visceral leishmaniasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Perirectal abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Malaria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 11 | 0 | 16 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 4 | 0 | 0 | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Bipolar disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Schizoaffective disorder (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alcoholism (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Conversion disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depression suicidal (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mood altered (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cardiomegaly (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram abnormal (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 5 | 0 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anastomotic leak (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Collapse of lung (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0/0 | 0
Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Penis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Paralysis (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myoclonus (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Post herpetic neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breast mass (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fibrocystic breast disease (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Breast enlargement (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anal stenosis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urethral disorder (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pterygium (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperthyroidism (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thyroiditis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FPV Population (APV30001) (N=119) | NFV Population (APV30001) (N=18) | FPV Population (APV30002) (N=221) | NFV Population (APV30002) (N=54) | FPV/RTV QD Population (APV30003) (N=73) | FPV/RTV BID Population (APV30003) (N=78) | PI-Naïve Population (Other Studies) (N=104) | PI-Experienced Population (Other Studies) (N=86) | Final Analysis Population (APV30005) (N=111)
Diarrhoea (Gastrointestinal disorders) | 51 | 5 | 131 | 15 | 27 | 37 | 16 | 14 | 14
Nausea (Gastrointestinal disorders) | 47 | 2 | 100 | 8 | 21 | 21 | 9 | 0 | 7
Upper respiratory tract infection (Infections and infestations) | 42 | 4 | 69 | 30 | 22 | 19 | 21 | 8 | 32
Nasopharyngitis (Infections and infestations) | 39 | 10 | 48 | 4 | 12 | 19 | 16 | 14 | 23
Rash (Skin and subcutaneous tissue disorders) | 35 | 2 | 41 | 7 | 8 | 12 | 4 | 1 | 7
Headache (Nervous system disorders) | 34 | 3 | 59 | 3 | 14 | 28 | 10 | 6 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 0 | 56 | 13 | 13 | 13 | 5 | 6 | 10
Fatigue (General disorders) | 22 | 1 | 54 | 4 | 18 | 17 | 6 | 4 | 3
Vomiting (Gastrointestinal disorders) | 20 | 2 | 53 | 7 | 17 | 9 | 4 | 3 | 4
Pyrexia (General disorders) | 19 | 0 | 30 | 3 | 8 | 6 | 6 | 8 | 1
Depression (Psychiatric disorders) | 18 | 0 | 30 | 6 | 13 | 18 | 10 | 9 | 6
Sinusitis (Infections and infestations) | 16 | 2 | 23 | 5 | 6 | 11 | 7 | 8 | 2
Bronchitis (Infections and infestations) | 15 | 0 | 40 | 9 | 13 | 8 | 9 | 10 | 8
Insomnia (Psychiatric disorders) | 15 | 0 | 32 | 5 | 13 | 15 | 9 | 4 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 0 | 29 | 7 | 11 | 11 | 5 | 2 | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14 | 0 | 17 | 5 | 10 | 7 | 5 | 3 | 7
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 14 | 1 | 18 | 0 | 5 | 9 | 3 | 6 | 0
Anogenital warts (Infections and infestations) | 13 | 0 | 5 | 2 | 9 | 1 | 4 | 3 | 1
Dizziness (Nervous system disorders) | 13 | 2 | 25 | 0 | 3 | 9 | 1 | 4 | 1
Gastroenteritis (Infections and infestations) | 13 | 2 | 14 | 8 | 7 | 5 | 6 | 3 | 4
Influenza (Infections and infestations) | 13 | 0 | 37 | 7 | 12 | 8 | 9 | 6 | 12
Herpes simplex (Infections and infestations) | 12 | 0 | 30 | 4 | 0 | 2 | 1 | 2 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 2 | 37 | 8 | 14 | 17 | 9 | 9 | 7
Abdominal pain (Gastrointestinal disorders) | 10 | 0 | 32 | 3 | 9 | 13 | 1 | 5 | 4
Pharyngitis (Infections and infestations) | 10 | 2 | 14 | 4 | 7 | 5 | 1 | 3 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 10 | 1 | 18 | 4 | 11 | 7 | 1 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 9 | 0 | 7 | 1 | 0 | 4 | 1 | 2 | 0
Anxiety (Psychiatric disorders) | 8 | 0 | 21 | 3 | 11 | 12 | 4 | 2 | 2
Asthenia (General disorders) | 8 | 1 | 11 | 1 | 3 | 7 | 3 | 2 | 0
Hypertension (Vascular disorders) | 8 | 0 | 20 | 1 | 3 | 5 | 5 | 1 | 11
Oedema peripheral (General disorders) | 8 | 0 | 10 | 2 | 1 | 3 | 1 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 12 | 6 | 2 | 2 | 2 | 2 | 9
Abdominal pain upper (Gastrointestinal disorders) | 7 | 0 | 20 | 3 | 7 | 4 | 1 | 4 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 0 | 9 | 1 | 3 | 2 | 6 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 7 | 1 | 16 | 0 | 8 | 6 | 5 | 4 | 2
Lipodystrophy acquired (Skin and subcutaneous tissue disorders) | 7 | 0 | 9 | 0 | 2 | 1 | 2 | 3 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 7 | 0 | 11 | 1 | 4 | 4 | 1 | 2 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 2 | 2 | 1 | 1 | 1 | 1 | 0
Chest discomfort (General disorders) | 6 | 0 | 4 | 0 | 0 | 1 | 0 | 0 | 0
Dermititis (Skin and subcutaneous tissue disorders) | 6 | 0 | 6 | 0 | 2 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 6 | 0 | 18 | 1 | 3 | 7 | 0 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 1 | 8 | 0 | 7 | 3 | 1 | 0 | 3
Paraesthesia (Nervous system disorders) | 6 | 1 | 10 | 0 | 8 | 6 | 0 | 2 | 1
Urinary tract infection (Infections and infestations) | 6 | 0 | 11 | 6 | 3 | 1 | 1 | 1 | 7
Dental caries (General disorders) | 0 | 2 | 1 | 1 | 1 | 1 | 0 | 0 | 2
Pneumonia (Infections and infestations) | 4 | 2 | 2 | 3 | 3 | 2 | 0 | 3 | 2
Vaginal infection (Infections and infestations) | 2 | 2 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Abscess limb (Infections and infestations) | 4 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Aphthous stomatitis (Gastrointestinal disorders) | 2 | 1 | 6 | 2 | 1 | 1 | 1 | 0 | 2
Bronchopneumonia (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Burns second degree (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 4 | 1 | 4 | 2 | 2 | 1 | 2 | 0 | 0
Conjunctivitis (Eye disorders) | 4 | 1 | 14 | 2 | 3 | 7 | 2 | 3 | 2
Constipation (Gastrointestinal disorders) | 2 | 1 | 8 | 3 | 4 | 4 | 2 | 4 | 2
Eczema (Skin and subcutaneous tissue disorders) | 5 | 1 | 5 | 2 | 1 | 3 | 0 | 0 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 5 | 1 | 14 | 4 | 1 | 0 | 3 | 3 | 1
Gastritis (Gastrointestinal disorders) | 5 | 1 | 2 | 1 | 3 | 1 | 2 | 1 | 4
Hot flush (Vascular disorders) | 0 | 1 | 4 | 0 | 0 | 1 | 2 | 0 | 2
Joint sprain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4 | 1 | 2 | 0 | 2 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 16 | 1 | 3 | 5 | 0 | 3 | 0
Parasitic infection intestinal (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pelvic inflammatory disease (Gastrointestinal disorders) | 4 | 1 | 3 | 0 | 0 | 1 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal candidiasis (Infections and infestations) | 0 | 1 | 6 | 1 | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 5 | 1 | 1 | 3 | 1 | 0 | 0
Vulvovaginitis trichomonal (Infections and infestations) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 5 | 1 | 18 | 7 | 3 | 6 | 4 | 1 | 7
Chest pain (General disorders) | 5 | 0 | 19 | 5 | 3 | 5 | 4 | 1 | 3
Paraesthesia oral (Nervous system disorders) | 1 | 0 | 19 | 0 | 7 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 4 | 0 | 18 | 1 | 2 | 3 | 2 | 2 | 3
Blood triglycerides increased (Investigations) | 2 | 0 | 17 | 1 | 3 | 3 | 2 | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 5 | 0 | 15 | 1 | 0 | 5 | 1 | 1 | 0
Hypoasthesia (Nervous system disorders) | 3 | 0 | 14 | 3 | 3 | 5 | 0 | 0 | 0
Sexual transmission of infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 14 | 5 | 2 | 0 | 2 | 0 | 2
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 13 | 0 | 2 | 7 | 2 | 1 | 2
Lipase increased (Investigations) | 3 | 0 | 13 | 0 | 6 | 2 | 0 | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 0 | 13 | 2 | 9 | 4 | 2 | 4 | 12
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 13 | 1 | 3 | 1 | 5 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 3 | 0 | 12 | 3 | 5 | 5 | 2 | 0 | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 12 | 3 | 3 | 5 | 1 | 1 | 2
Seasonal allergy (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 12 | 0 | 2 | 1 | 2 | 0 | 2
Alanine aminotransferase increased (Investigations) | 4 | 0 | 10 | 4 | 4 | 2 | 0 | 4 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 7 | 4 | 7 | 5 | 0 | 1 | 0
Ear infection (Infections and infestations) | 2 | 0 | 0 | 3 | 3 | 1 | 1 | 1 | 0
Syphilis (Infections and infestations) | 5 | 0 | 5 | 3 | 1 | 1 | 4 | 2 | 0
Tonsillitis (Infections and infestations) | 5 | 0 | 6 | 3 | 0 | 1 | 1 | 0 | 1
Viral infection (Infections and infestations) | 1 | 0 | 7 | 3 | 1 | 1 | 4 | 0 | 0
Skin papilloma (Skin and subcutaneous tissue disorders) | 0 | 0 | 5 | 1 | 10 | 4 | 1 | 2 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 3 | 0 | 9 | 1 | 6 | 6 | 2 | 2 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 4 | 0 | 3 | 7 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 5 | 0 | 5 | 3 | 1 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 0 | 6 | 0 | 3 | 5 | 5 | 0 | 1
Influenza like illness (General disorders) | 2 | 0 | 6 | 1 | 3 | 5 | 0 | 2 | 0
Tinea pedis (Infections and infestations) | 5 | 0 | 9 | 2 | 0 | 2 | 6 | 0 | 3
Respiratory tract infection viral (Infections and infestations) | 0 | 0 | 4 | 2 | 4 | 3 | 3 | 0 | 10
Rhinitis (Infections and infestations) | 2 | 0 | 7 | 2 | 0 | 0 | 0 | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.